CLINICAL TRIAL: NCT06410378
Title: Ultrasound-Guided Erector Spinae Block Versus Serratus Anterior Block for Perioperative Analgesia In Patients Undergoing Modified Radical Mastectomy Surgery
Brief Title: s Serratus Anterior Block for Perioperative Analgesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Asmaa Mohammed Galal El-Deen, lecture of anesthesia and ICU, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZagazigS
Record Dates: First submitted 2024-03-18; First posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Mastectomy; Postoperative Pain
Keywords: Erector Spinae Block; Serratus anterior Block; Perioperative Analgesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: The patients will be divided randomly by a computer-generated randomization table into three equal groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Erector Spinae Plane Block (Active Comparator): patient place in sitting position. Type of needle Using 22-gauge spinal needle 10 cm Linear ultrasound probe is placed in a longitudinal parasagittal orientation 3 cm lateral to the T5 spinous process.
  The erector spinae muscle is identified superficial to the tip of The T5 transverse process.
  Needle insertion The needle is inserted in- plane superior to inferior approach. The tip of the needle is placed into the fascial plane on the deep aspect of erector spinae muscle.
  The location of the needle tip is confirmed by visible normal saline fluid spread separating erector spinae muscle off the bony shadow of the transverse process on ultrasonographic imaging .
  Local anesthetic and volume Injection of 20 ml of bupivacaine 0.25 %.
  Interventions: Procedure: Erector Spinae Plane Block
- Serratus Anterior Plane Block: (Active Comparator): The patient lies supine with placing the ipsi-lateral upper limb in abduction at 90° positio Using 22-gauge spinal needle 10 cm length. After skin sterilization, Ultrasound device with high frequency [9-12] and superficial linear probe that is first placed inferior to the middle of the clavicle and moved laterally and downward to locate the 1st rib where pectoralis major and pectoralis minor muscles are identified at this US window.
  The US probe is moved toward axilla till serratus anterior muscle is identified above 2nd, 3rd and 4th ribs. The transducer is held at a slightly oblique angle at the level of the 4th and 5th rib, with the upper edge supero-anterior and the lower edge infero-anterior.
  Needle insertion After infiltration of the skin at puncture site with 3 ml of lidocaine 1%, the needle is inserted inplane between the anterior serratus and the latissimus dorsi muscle on the mid-axillary line.
  Injection of 20 mL of 0.25% bupivacaine.
  Interventions: Procedure: Serratus Anterior Plane Block
- control group (Active Comparator): patients will receive only general anesthesia for Modified Radical Mastectomy.
  Interventions: Procedure: controll group

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — Patient will receive 20 ml of bupivacaine 0.25 % through Erector Spinae Plane Block approach
  Other Names: Group E
  Arms: Erector Spinae Plane Block
Procedure: Serratus Anterior Plane Block — Patient will receive 20 ml of bupivacaine 0.25 % through Serratus Anterior Plane Block approach.
  Other Names: Group S
  Arms: Serratus Anterior Plane Block:
Procedure: controll group — patient will receive general anesthesia
  Other Names: Group C
  Arms: control group

SUMMARY:
Modified radical mastectomy is one of the commonly performed breast surgery. Postoperative pain following mastectomy should be minimised, as in a number of women it may chronically persist for months in the form of postmastectomy pain syndrome.

Morphine administration for acute pain after mastectomy surgery has many side effects. Regional block techniques as paravertebral block and thoracic epidural anathesia has possible complications and technical difficulties.

The new alternative regional techniques such as erector spinae plane block and serratus anterior plane block are clinical trials for providing a safe, easy and painless anesthetic procedure with good hemodynamic and recovery profile with adequate perioperative analgesia for a large section of patients undergoing mastectomy operation in order to reduce opiods consumption and subsequently avoid opiod-related adverse effects.

DETAILED DESCRIPTION:
Breast cancer is the most common malignancy of women all over the world. Unfortunately, two-thirds of women who undergo breast cancer surgery are reported to develop chronic pain in the postoperative period. Surgery type, radiation therapy, and clinically acute pain are the most important risk factors for the development of more intense chronic pain.

With improved diagnostic techniques and treatment regimens, prognosis in breast cancer is improving, with the 5-year survival of patients diagnosed with primary breast cancer having increased to approximately 85%. Persistent post-surgical pain states in this group is reported in 30-50% of patients, up to half of whom may have pain well beyond 5 years. Over one-third of patients who underwent breast cancer surgery have inadequately controlled acute post-operative pain.

There are several ways to manage pain after mastectomy. Common systemic medications, particularly opioids, have different side effects, such as itching, nausea, vomiting and respiratory depression. Non-steroidal anti-inflammatory drugs are associated with impaired renal function and hemorrhagic disorders.

Regional anesthesia has been believed as one of the formats for effective perioperative pain control. Regional blocks using ultrasound-guide has become a perfect supplement to general anesthesia for extending analgesia after modified radical mastectomy. The advantage includes post-operative pain relief prolongation, a decrease in analgesic requirement post-operatively, a reduction in nausea and vomiting scores and probability for ambulatory discharge and hospital stay.

The complex innervation of breast tissues poses a great challenge for the anesthesiologists to provide adequate perioperative analgesia by ultrasound guided regional blocks. Thoracic epidural, interscalene brachial plexus block, paravertebral block, pectoral nerve I and pectoral nerve II blocks have been used in different studies with good results. There are also technically simple regional blocks as ultrasound-guided Serratus anterior Plane (US-guided SAP) block and erector spinae plane (US-guided ESP) block which can be used effectively for this purpose.

Forero et al. described ultrasound-guided Erector Spinae Plane (US-ESP) block as a novel analgesic technique in which local anesthetic injection is done beneath the erector spinae muscle. Previous studies reported effective postoperative pain reduction with ESP block after radical mastectomy surgery. Nevertheless, few studies have compared the efficacy of ESP block with another block technique.

The Serratus Anterior Plane block (SAP) provides anterolateral and partial posterior thoracic wall analgesia, affecting dermatomes from T2 to T9. SAP is affecting predominantly the lateral cutaneous branches of the thoracic intercostal nerves, along with intercostobrachial, thoracodorsal and long thoracic nerves. The block is performed further posteriorly and caudally than Pectoral Nerve Block-2, where the target nerves are located between the serratus anterior and the latissimus dorsi muscles.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from the patient.

  * Age: 21 - 60 years old.
  * Gender: female patients.
  * Body mass index: < 35 kg/m2.
  * Physical status: ASA grade I-II (American society of anesthiologists).
  * Type of operation: unilateral modified radical mastectomy operation.

Exclusion Criteria:

* • Patient with known history of allergy to study drugs.

  * Chronic use of analgesics or drug dependence.
  * Patients not able to understand pain assessment test.
  * Anatomical abnormalities.
  * Neuropathic disease.
  * Pregnancy or breast feeding.
  * Other contraindication of regional anesthesia e.g. septic focus at site of injection.
  * patient with coagulopathy or on anticoagulant therapy.

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-05-10 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
time of first analgesia requirement | during 24 hours postoperative
  first time patient asks rescue analgesia and total morphine consumption post-operative.

SECONDARY OUTCOMES:
onset of Sensory block. | within 20 minutes after block
  time needed for onset of sensory block.
assessment of sensory block | within 8 hours after giving block
  quality and duration of block

OTHER OUTCOMES:
dynamic pain scores | at 2 hours, 4 hours, 8 hours, 12 hours, 18 hours and 24 hours post-operatively.
  Visual analog scale (VAS) of 0-10, where 0= No pain and 10= Maximum worst pain.
Static pain scores | at 2 hours, 4 hours, 8 hours, 12 hours, 18 hours and 24 hours post-operatively.
  Visual analog scale (VAS) of 0-10, where 0= No pain and 10= Maximum worst pain.

CONTACTS AND LOCATIONS:
Overall Officials: Halah I Zanfaly, MD, Principal Investigator — Zagazig University
Locations (1):
- Zagazig, Zagazig, MD, Egypt

IPD SHARING:
Plan to Share IPD: Yes
planned after the completion of the study and publication
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: planned after the completion of the study and publication
Access Criteria: principal investigator

REFERENCES:
- [Background] Altiparmak B, Korkmaz Toker M, Uysal AI, Turan M, Gumus Demirbilek S. Comparison of the effects of modified pectoral nerve block and erector spinae plane block on postoperative opioid consumption and pain scores of patients after radical mastectomy surgery: A prospective, randomized, controlled trial. J Clin Anesth. 2019 May;54:61-65. doi: 10.1016/j.jclinane.2018.10.040. Epub 2018 Nov 3. PMID 30396100
- [Background] Blanco R, Parras T, McDonnell JG, Prats-Galino A. Serratus plane block: a novel ultrasound-guided thoracic wall nerve block. Anaesthesia. 2013 Nov;68(11):1107-13. doi: 10.1111/anae.12344. Epub 2013 Aug 7. PMID 23923989
- [Background] Eldemrdash AM, Abdelzaam EM: By Ultrasonic-Guided Erector Spinae Block, Thoracic Paravertebral Block versus Serratus Anterior Plane Block by Articaine with Adrenaline during Breast Surgery with General Anesthesia: A Comparative Study of Analgesic Effect Post-Operatively: Double Blind Randomized, Controlled Trial, Open Journal of Anesthesiology 2019; 9: 68-82.
- [Background] FitzGerald S, Odor PM, Barron A, Pawa A. Breast surgery and regional anaesthesia. Best Pract Res Clin Anaesthesiol. 2019 Mar;33(1):95-110. doi: 10.1016/j.bpa.2019.03.003. Epub 2019 Apr 6. PMID 31272657
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Gad M, Abdelwahab K, Abdallah A, Abdelkhalek M, Abdelaziz M. Ultrasound-Guided Erector Spinae Plane Block Compared to Modified Pectoral Plane Block for Modified Radical Mastectomy Operations. Anesth Essays Res. 2019 Apr-Jun;13(2):334-339. doi: 10.4103/aer.AER_77_19. PMID 31198256
- [Background] Khemka R, Chakraborty A. Ultrasound-guided modified serratus anterior plane block for perioperative analgesia in breast oncoplastic surgery: A case series. Indian J Anaesth. 2019 Mar;63(3):231-234. doi: 10.4103/ija.IJA_752_18. PMID 30988539
- [Background] Metwally AA, Elfeky EM, Abo Elenain KM, Yousef IM: Scoring systems in Anesthesia. Nature and Science 2016; 14: 47-48.
- [Background] Rahimzadeh P, Imani F, Faiz SHR, Boroujeni BV. Impact of the Ultrasound-Guided Serratus Anterior Plane Block on Post-Mastectomy Pain: A Randomised Clinical Study. Turk J Anaesthesiol Reanim. 2018 Sep;46(5):388-392. doi: 10.5152/TJAR.2018.86719. Epub 2018 Sep 4. PMID 30263863
- [Background] Ross VH, Pan PH, Owen MD, Seid MH, Harris L, Clyne B, Voltaire M, Eisenach JC. Neostigmine decreases bupivacaine use by patient-controlled epidural analgesia during labor: a randomized controlled study. Anesth Analg. 2009 Aug;109(2):524-31. doi: 10.1213/ane.0b013e31819518e4. Epub 2009 Apr 17. PMID 19377050
- [Background] Singh S, Kumar G, Akhileshwar. Ultrasound-guided erector spinae plane block for postoperative analgesia in modified radical mastectomy: A randomised control study. Indian J Anaesth. 2019 Mar;63(3):200-204. doi: 10.4103/ija.IJA_758_18. PMID 30988534
- [Background] Swami SS, Keniya VM, Ladi SD, Rao R. Comparison of dexmedetomidine and clonidine (alpha2 agonist drugs) as an adjuvant to local anaesthesia in supraclavicular brachial plexus block: A randomised double-blind prospective study. Indian J Anaesth. 2012 May;56(3):243-9. doi: 10.4103/0019-5049.98767. PMID 22923822

DOCUMENTS (1):
  • Study Protocol (2024-04-20): https://cdn.clinicaltrials.gov/large-docs/78/NCT06410378/Prot_000.pdf